CLINICAL TRIAL: NCT06754644
Title: A Randomized, Double-blind, Multicenter Phase III Clinical Study to Compare the Efficacy and Safety of QL2107 Versus Keytruda® in Combination With Chemotherapy in the Treatment of Metastatic Non-squamous Non-small-cell Lung Cancer
Brief Title: A Study to Evaluate Efficacy, and Safety of QL2107 Plus Chemo and Compare With Keytruda in Participants With IV nqNSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2107-301-CN
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-12

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Carboplatin; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2107 (Experimental)
  Interventions: Drug: QL2107; Drug: Pemetrexed; Drug: Carboplatin
- Keytruda® (Active Comparator)
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Keytruda®

INTERVENTIONS:
Drug: QL2107 — 200mg on day 1 of each 21-day cycle of the study
  Arms: QL2107
Drug: Pemetrexed — 500 mg/m2 on Day 1 of each 21-day cycle of the study
Drug: Carboplatin — Target AUC of 5 mg/mL/min on Day 1 of each 21-day cycle up to 4 cycles
Drug: Keytruda® — 200mg on day 1 of each 21-day cycle of the study
  Arms: Keytruda®

SUMMARY:
The goal of this clinical trial is to compare the efficacy similarities between QL2107 and Keytruda in metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily participate, sign the Informed Consent Form (ICF), and are able to comply with the study procedures;
* Subjects aged ≥ 18 and ≤ 75 years at enrollment, male or female;
* Histologically or cytologically confirmed metastatic (stage IV) non-squamous NSCLC as per the American Joint Committee on Cancer (AJCC) 8th Edition; if multiple tumor histologies are present, the predominant cell type should be classified;
* No EGFR sensitive mutations or ALK gene translocations.
* Expected survival ≥ 3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0 or 1;

Exclusion Criteria:

* Pulmonary radiation therapy > 30 Gy within 6 months prior to the first dose;
* Palliative radiation therapy completed within 7 days prior to the first dose;
* Any other form of anti-tumor therapy expected to be required during the study;
* Uncontrolled or symptomatic pericardial effusion, pleural effusion and ascites requiring repeated paracentesis and drainage;
* Presence of metastases to brain stem, meninges and spinal cord or compression;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
clinical equivalence | 24-week
  The 24-week objective response rate (24-week ORR, defined as the proportion of subjects who achieve CR or PR based on best efficacy at any time within 24 weeks after administration, evaluated according to RECIST 1.1) assessed by the Independent Review Committee (IRC)

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University Cancer Hospital, Jinan, Shandong, China